CLINICAL TRIAL: NCT07137403
Title: Unsteady Gait in Older People May be a Common and Treatable Neurological Disease Associated With Increased Mortality - Damage to the Glymphatic System May be the Cause
Brief Title: Unsteady Gait in Older People May be a Common and Treatable Neurological Disease Associated With Increased Mortality
Acronym: VESPR2
Status: Enrolling by invitation | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government); The Swedish Brain Foundation (Hjärnfonden) (Unknown)
Responsible Party: Principal Investigator, Jenny Ma Larsson, Researcher, Umeå University
Other Study IDs: 2025-02534-01
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH); Gait Disorders, Neurologic; Gait Disorders in Old Age
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Higher-level gait disorder: Individuals who in our previous study had a higher-level gait disorder
- Other gait disorder/No gait disorder: Individuals who did not have a higher-level gait disorder during their visit in our pervious study

SUMMARY:
We live in an aging population and a third of the older population has a gait disorder that may cause institutionalization, and increased mortality. Sixteen percent of them have a slow, unsteady, neurological gait disorder, called Higher-Level Gait Disorder (HLGD). A known cause of HLGD is Idiopathic Normal Pressure Hydrocephalus (INPH), which is a treatable neurological disease. More than half of individuals with HLGD meet the diagnostic criteria for INPH as they have wide brain ventricles on MRI images of the brain, but far from all of these are in contact with the healthcare system. Possibly, HLGD without wide brain ventricles and where no other known explanation for the symptom is found could be a variant of or a precursor to INPH.

Gait disorder is common among older people and can lead to falls and reduced quality of life. Complications after falls contribute to both increased mortality and increased costs in society. Therefore, it is important to have a solid knowledge of different types of gait disorders and how they can be treated. Our research will contribute with information about how HLGD affects the individual and how affected individuals can be investigated and helped.

The disease mechanisms behind INPH and often behind HLGD are unknown. It is also unknown how often older individuals are affected by HLGD and how high the mortality is for those affected. It is likely that the incidence of HLGD is high and that it is linked to an increased mortality. It is also likely that the disease mechanism behind the symptom is the same as that of INPH and that HLGD can be detected with the help of brain imaging.

In this epidemiological cohort study, we want to answer the following overarching questions:

What is the incidence and mortality of HLGD and INPH? Can HLGD be predicted using biomarkers and what disease mechanism causes HLGD?

ELIGIBILITY:
Inclusion Criteria:

* Participation in the study "Ventriculomegaly and gait disturbance in the senior population in the Region of Västerbotten" (VeSPR)

Exclusion Criteria:

* Bedridden
* Inability to leave informed consent due to cognitive decline

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: In the VeSPR study, a questionnaire about gait problems was sent to 6467 randomly selected individuals aged 65-84 years in Umeå. All with self-perceived gait problems (n=1510) and 513 controls without self-perceived gait problems were invited to a physical examination by a physician as well as clinical examinations of gait and balance, cognition and comorbidity. Of these, 1047 participated in clinical examinations (798 with gait disorders and 249 controls), 909 of them had a subsequent MRI of the brain and 98 had a computed tomography (CT) scan. With a theoretical constant mortality rate of 2.3%/year (Swedish official statistics on mortality in the age-group), there is a remaining population of 910 individuals from the previous study to invite to the 6-year follow-up. We expect about half of these will choose to participate, resulting in approximately 450 participants.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 years
6 year incidence of Higher-Level Gait Disorder and Idiopathic Normal Pressure Hydrocephalus | 6 years
  Number of individuals that have developed a Higher-Level Gait Disorder and Idiopathic Normal Pressure Hydrocephalus since their last visit to us, in our previous study VESPR.

SECONDARY OUTCOMES:
MRI Biomarkers for prediction of HLGD | 6 years
  MRI biomarkers commonly used in hydrocephalus diagnostics such as Evans Index, Callosal Angle and DESH will be evaluated for prediction of HLGD development. New biomarkers will also be investigated as potential new diagnostic tools.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Larsson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No